CLINICAL TRIAL: NCT02056275
Title: A Study of an Oral Nutrition Supplement (ONS) in Children.
Status: Completed | Phase: Not Applicable | Type: Interventional
Sponsor: Abbott Nutrition (Industry)
Responsible Party: Sponsor
Allocation: Randomized | Model: Parallel | Masking: None
Other Study IDs: DA01
Record Dates: First submitted 2014-02-04; First posted 2014-02-05 (Estimated); Last update posted 2015-03-06 (Estimated); Status verified 2014-10

CONDITIONS: Growth
MeSH Terms: interventions — Nutrition Assessment

STUDY DESIGN:
Oversight: Data Monitoring Committee: No

ARMS (2):
- ONS + dietary counseling (Experimental): ONS/day + dietary counseling
  Interventions: Other: Nutrition supplement + dietary counseling
- Dietary counseling (Active Comparator): Dietary counseling
  Interventions: Other: Dietary Counseling

INTERVENTIONS:
Other: Nutrition supplement + dietary counseling — Nutritionally balanced nutritional supplement providing 1.0 kcal/ml.
  Other Names: Commercially available nutritional supplement.
  Arms: ONS + dietary counseling
Other: Dietary Counseling — Dietary counseling provided at each study visit by study dietitian.
  Arms: Dietary counseling

SUMMARY:
To assess the effect of oral nutritional supplementation with dietary counseling versus dietary counseling alone on growth of preschool children over a period of 90 days.

ELIGIBILITY:
Inclusion Criteria:

1. Age of 24-72 months (inclusive), both genders.
2. Diagnosed with current acute upper respiratory tract infection.
3. Weight-for-age between 3rd - 15th percentile according to WHO Growth Charts.
4. Identified as a picky eater.
5. Able to consume foods and beverages orally.
6. Willing to abstain from additional non-study provided protein supplements or nutritional supplements throughout the study period.

Exclusion Criteria:

1. Current illness requiring hospitalization.
2. Gastrointestinal infection and/or acute diarrhea at the time of inclusion in the study.
3. Currently taking medication that could affect absorption/metabolism of study product or weight of the child.
4. Diagnosed with recurrent respiratory infections due to cystic fibrosis, immunodeficiency syndromes, and congenital abnormalities of the respiratory tract, congenital lung and ciliary abnormalities, an unsuspected foreign body and asthma.
5. Active tuberculosis, acute hepatitis B or C, or HIV, malignancy.
6. History of diabetes mellitus.
7. Received antibiotic therapy within the last two weeks before start of the study.
8. Dysphagia, aspiration risk, difficulty in swallowing due to acquired / congenital abnormalities that would hamper oral intake of the study product.
9. Clinically significant nutritional deficiency requiring specific treatment with any other nutritional supplement (not study product).

Ages: 24 Months to 72 Months | Sex: All | Healthy Volunteers: No
Age Groups: Child
Enrollment: 256 (Actual)
Dates: Start 2013-08; Primary Completion 2014-04 (Actual); Study Completion 2014-04 (Actual)

PRIMARY OUTCOMES:
Weight | Study Day (SD) 1 to 90
  Change in weight-for-age from Day 1 to Day 90

SECONDARY OUTCOMES:
Respiratory Infections | Study Day (SD) 1 to 90
  Number and duration of recurrent acute upper respiratory tract infections per month during the study period.
Sick Days | Study Day (SD) 1 to 90
  Number of sick days per month assessed by the presence of any acute upper respiratory tract infections during the study period.
Doctor Visits | Study Day (SD) 1 to 90
  Number of unscheduled visits per month due to development of acute upper respiratory tract infections during the study period.
Dietary Intake | Study Day (SD) 1 to 90
  Average energy consumption (values and changes from baseline).
Appetite Score | Study Day (SD) 3, 10, 30, 60 and 90
  Change in appetite score (values and changes from baseline)

CONTACTS AND LOCATIONS:
Overall Officials: Vinita Satyavrat, MD, Study Chair — Abbott Nutrition
Locations (8):
- India (8):
  - St. Theresa's Hospital, Hyderabad, Andhra Pradesh
  - Praveen Cardiac Centre, Vijayawada, Andhra Pradesh
  - Sangini Hospital, Ahmedabad, Gujarat
  - Kasturba Medical College and Hospital, Manipal, Karnataka
  - Noble Hospital, Pune, Maharashtra
  - TN Medical College & BYL Nair Hospital, Mumbai, Mumbai
  - Seth GS Medical College and KEM Hospital, Mumbai-12, Mumbai
  - Institute of Child Health, Kolkata, West Bengal